CLINICAL TRIAL: NCT05509725
Title: Efficacy and Safety of a Probiotic Formulation in Adults With Irritable Bowel Syndrome With Diarrhea (IBS-D): A Multicenter, Randomized, Prospective, Placebo-Controlled, Double-Blind, Phase IV Clinical Study
Brief Title: Efficacy and Safety of a Probiotic Formulation in Adults With Irritable Bowel Syndrome With Diarrhea (IBS-D)
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Lallemand Health Solutions (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: C-005
Record Dates: First submitted 2022-07-01; First posted 2022-08-22 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: IBS - Irritable Bowel Syndrome
Keywords: IBS-D; Probiotics
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants in this group will be randomized to receive probiotic formulation for the following 8 weeks.
  Interventions: Drug: Probiotic formulation
- Control (Placebo Comparator): Participants in this group will be randomized to receive placebo for the following 8 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Probiotic formulation — Participants will be asked to take 2 doses daily
  Arms: Intervention
Drug: Placebo — Participants will be asked to take 2 doses daily
  Arms: Control

SUMMARY:
The purpose of the study is to monitor safety and to evaluate the efficacy of a probiotic formulation on abdominal pain, abnormal defecation, comorbid mood disorders (anxiety and depression) as well as general quality of life in adults with IBS-D.

DETAILED DESCRIPTION:
To monitor safety and to evaluate the efficacy of a probiotic formulation on severity of gastrointestinal symptoms (abdominal pain, abnormal defecation), anxiety, depression and quality of life in adult participants with IBS-D.

ELIGIBILITY:
Inclusion Criteria:

* Experiencing symptoms of IBS-D
* Having a diagnosis of IBS-D based on Rome IV criteria
* Participants with symptom onset at least 6 months before diagnosis
* Having a normal colonoscopy result in their medical file

Exclusion Criteria:

* A history of inflammatory or immune-mediated gastrointestinal diseases
* Diagnosed with a co-existing organic gastrointestinal disease which can affect the study
* Currently undergoing a treatment for other severe conditions such as coronary disease, neurological disorder, kidney or liver disease,
* Currently diagnosed with an eating disorder,
* Having undergone any abdominal surgery including cholecystectomy, with the exception of hernia repair or appendectomy
* Currently diagnosed with any mood- or anxiety-related disorder, major psychiatric illness, or participants with a history of suicidal ideation, or current suicidal ideation,
* Regular use of anti-diarrhea medications and laxatives however occasional use is permitted (≤ than once a month); if current use is > once per month a one month wash out is needed,
* Unwilling to avoid the use of antidiarrheal or laxative medication on an "as-needed basis" during the full length of the study,
* Pregnant, breast-feeding or planning on becoming pregnant.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2022-08-11 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Change in Abdominal Pain | 8 weeks
  Change in abdominal pain intensity using Visual Analog Scale (VAS) from 0 (no symptom) to 10 (worst possible)
Change in Defecation consistency | 8 weeks
  Change in abnormal defecation consistency using the Bristol Stool Scale (BSS) from Type 1 (severe constipation) to Type 7 (severe diarrhea)

SECONDARY OUTCOMES:
Change Abdominal pain intensity | up to 10 weeks
  Change in abdominal pain intensity using Visual Analog Scale (VAS) from 0 (no symptom) to 10 (worst possible)
Abnormal defecation consistency | up to 10 weeks
  Change in abnormal defecation consistency using the Bristol Stool Scale (BSS) from Type 1 (severe constipation) to Type 7 (severe diarrhea)
Stool frequency | up to 10 weeks
  Measured as the average number of stools per week
Abdominal discomfort | up to 10 weeks
  Using questionnaire in participants diary
Perceived Stress | 8 weeks
  Using the Perceived Stress Scale (PSS) grading from 0 (low stress) to 40 (high perceived stress)
Change in Irritable Bowel Syndrome Symptom Severity Scores | 8 weeks
  Using the The irritable bowel severity scoring system (IBS-SSS)

CONTACTS AND LOCATIONS:
Overall Officials: Serhat Bor, Prof. Dr., Principal Investigator — Ege University
Locations (1):
- Ege University Faculty of Medicine, Gastroenterology Department, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
After publications of the results, de-identified data will be shared with qualified researchers and scientists upon reasonable request to the sponsor including a detailed proposal of the intended use of the data, as per the Lallemand Health Solutions Inc. Policy on Clinical Trial Transparency and Data Sharing (available upon request).